CLINICAL TRIAL: NCT01851434
Title: Natural History of Optic Neuritis
Status: Terminated | Type: Observational
Why Stopped: The original analyses could not be performed due to data inconsistencies across the study sites.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130104; 13-N-0104
Record Dates: First submitted 2013-05-09; First posted 2013-05-10 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: OCT; Multiple Sclerosis; Optic Neuritis; Magnetic Resonance Imaging (MRI); Natural History
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- healthy volunteers: age- and sex-matched to the participants with unilateral optic neuritis and a brain MRI suggestive of MS
- Patients with unilateral optic neuritis: Recruitment will proceed until 10 participants with a brain MRI suggestive of MS (obtained at any time point during the study) have completed the study.

SUMMARY:
Background:

- Optic neuritis often is a symptom of multiple sclerosis (MS). Many people who experience optic neuritis are later diagnosed with MS. MS disease activity seen on magnetic resonance imaging (MRI) scans is often greater than that seen in tests given during regular doctor's visits. Even though MRI is a helpful tool for studying optic neuritis and MS, more information is needed on how MS symptoms show up on MRI scans. Researchers want to use MRI scans to track changes in the optic nerve after an optic neuritis episode. This approach will help them study the relationship between optic neuritis and MS.

Objectives:

- To collect more information about the relationship between optic neuritis and multiple sclerosis.

Eligibility:

* Individuals between 18 and 50 years of age who have new optic neuritis.
* Individuals between 18 and 50 years of age who have new symptoms of MS other than optic neuritis.
* Healthy volunteers between 18 and 50 years of age.

Design:

* Participants will be screened with a physical exam and medical history. They may provide blood or urine samples.
* Participants with optic neuritis or other MS symptoms will have a baseline study visit. They will have a physical exam and full eye exam. To look for signs of MS, they will have evoked potential tests to see how the body responds to stimulation. They will also have an MRI scan to study any changes in the brain and optic nerves.
* After the first visit, participants will have steroid treatment for 5 days for the optic neuritis.
* Additional study visits will be given 1, 3, 6, 9, and 12 months after the baseline visit. The tests from the first visit, including the MRI scans, will be repeated at these visits.
* Healthy volunteers will have a baseline study visit. They will have a physical exam and full eye exam. They will have evoked potential tests to see how the body responds to stimulation. They will also have an MRI scan to study any changes in the brain and optic nerves.
* Healthy volunteers will have additional study visits 2 and 11 months after the baseline visit. The tests from the first visit, including the MRI scans, will be repeated at these visits.

DETAILED DESCRIPTION:
Objective

The goals of this pilot study are:

1. To assess the degree to which subacute changes in clinical, electrophysiological, and imaging measures can robustly predict retinal neuronal loss 12 months after acute optic neuritis.
2. To construct a composite score that integrates these subacute changes, can itself robustly predict retinal neuronal loss 12 months after acute optic neuritis, can be validated in future trials, and is likely to be modulated by drugs that promote tissue repair and neuroprotection in multiple sclerosis (MS).
3. To evaluate the usefulness of specialized magnetic resonance imaging (MRI) measures of the optic nerve in future clinical trials of drugs designed to promote tissue repair and neuroprotection. The primary hypothesis of the study is that peripapillary retinal nerve fiber layer (RNFL) thickness, which is generally agreed to reflect the integrity of optic nerve axons following optic neuritis, and which can be measured using spectral-domain optical coherence tomography (OCT) in the affected eye 12 months following optic neuritis, can be robustly predicted by changes in RNFL thickness between 1 and 3 months following symptom onset.

Study Population

The following cohorts will be recruited at each of the three study sites:

* Up to 30 participants with acute optic neuritis.
* Up to 15 healthy volunteers who are group-wise age- and sex-matched to the participants with unilateral optic neuritis.

Design

This is a one-year, prospective, multi-cohort, multi-site, pilot natural history study. Data obtained at NIH will be compared and aggregated with data obtained at other study sites, specifically the University of Utah-Moran Eye Center (in Salt Lake City) and Hebrew University-Hadassah Medical Center (in Jerusalem, Israel). Data will be gathered at baseline (optional) and at 1, 3, 6, 9, and 12 months in the patient cohort, and at 1, 3, and 12 months in the healthy volunteers.

Outcome Measures

The primary outcome measure is the RNFL thickness in the affected eye 12 months after optic neuritis.

Secondary outcome measures, all measured at 12 months, include:

* Measures of optic nerve structure: mean cross-sectional optic-nerve area; mean, parallel, and perpendicular diffusivity; and MTR all within the optic nerve lesion as visualized at baseline.
* Measures of brain structure: ventricular volume; T2 lesion volume along the visual pathway both sides considered together.
* Measures of retinal structure: ganglion cell layer + inner plexiform layer thickness in the affected eye.
* Measures of visual function: low-contrast letter acuity; high-contrast letter acuity; Pelli-Robson contrast sensitivity; object-from-motion detection; visual fields; and critical flicker-fusion frequency all in the affected eye.
* Measures of visual physiology: VEP amplitude; VEP latency all in the effected eye.

ELIGIBILITY:
* INCLUSION CRITERIA:

COHORT 1: Unilateral optic neuritis.

* Typical demyelinating optic neuritis based on the best clinical judgment of the investigators.
* Symptom onset within 46 weeks of enrollment OR patients with history of optic neuritis who were followed from symptom onset under a Neuroimmunology Branch natural history or screening protocol.
* For women of childbearing potential, willing to use acceptable forms of contraception (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods (condom or diaphragm) with spermicide or they have undergone surgical sterilization (hysterectomy, tubal ligation, or vasectomy in a partner) for the study duration.
* Able to provide informed consent.
* Willing and able to participate in all aspects of the trial.

COHORT 2: Healthy volunteers.

* No medical history that would interfere with study result interpretation, in the best clinical judgment of the investigators.
* Age greater than or equal to 18 years and less than or equal to 50 years.
* Able to provide informed consent.
* Willing and able to participate in all aspects of the trial.

EXCLUSION CRITERIA:

* History of signs or symptoms suspicious for MS, in the best clinical judgment of the investigators.
* Pateints-Disease-modifying therapy for MS prior to the onset of the current episode of optic neuritis (excludes oral or intravenous glucocorticoids: Healthy Volunteers - Previous or current use of disease-modifying therapy for MS (excluding oral or intravenous glucocorticoids.
* Previous history of clinical optic neuritis or a systemic disease associated with optic neuritis (e.g. sarcoidosis, lymphoma).
* Current or prior optic neuropathy (e.g. trauma, ischemia, glaucoma, optic nerve drusen).
* Previous history of a retinal disease (e.g. diabetic retinopathy, retinal drusen) other than uveitis.
* Previous history of an ophthalmic disease that in the best judgment of the investigator could affect ophthalmic imaging results.
* Previous history of a systemic disease that may mimic MS (e.g. neurosyphilis, neurosarcoidosis, CNS ymphoma, Si(SqrRoot)(Delta)gren s syndrome).
* Previous history of a systemic disease that in the best judgment of the investigator could confound study outcome.
* Current use of a TNF-alpha inhibitor (e.g. etanercept).
* Habitual use of illicit drugs that in the best judgment of the investigators could confound study outcome.
* Pregnant or breast-feeding.
* Unwilling to co-enroll on a Neuroimmunology Branch natural history or screening protocol currently 89-N-0045.
* Contraindication to MRI scanning.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Up to 30 participants with unilateral optic neuritis. Recruitment will proceed until 10 participants with a brain MRI suggestive of MS (obtained at any time point during the study) have completed the study. - Up to 15 healthy volunteers, age- and sex-matched to the participants with unilateral optic neuritis and a brain MRI suggestive of MS.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the RNFL thickness in the affected eye 12 months after optic neuritis | 12 months after optic neuritis
  RNFL thickness in the affected eye 12 months after optic neuritis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (3):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Utah, Salt Lake City, Utah
- Hadassah Hospital/Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Leaney J, Klistorner A, Arvind H, Graham SL. Dichoptic suppression of mfVEP amplitude: effect of retinal eccentricity and simulated unilateral visual impairment. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6549-55. doi: 10.1167/iovs.10-5769. Epub 2010 Jul 29. PMID 20671270
- [Background] Klistorner A, Arvind H, Garrick R, Yiannikas C, Paine M, Graham SL. Remyelination of optic nerve lesions: spatial and temporal factors. Mult Scler. 2010 Jul;16(7):786-95. doi: 10.1177/1352458510371408. Epub 2010 Jun 7. PMID 20530125
- [Background] Klistorner A, Arvind H, Garrick R, Graham SL, Paine M, Yiannikas C. Interrelationship of optical coherence tomography and multifocal visual-evoked potentials after optic neuritis. Invest Ophthalmol Vis Sci. 2010 May;51(5):2770-7. doi: 10.1167/iovs.09-4577. Epub 2009 Dec 30. PMID 20042660
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-N-0104.html